CLINICAL TRIAL: NCT06016335
Title: Artificial Intelligence Driven Synthetic CT to Substitute CT Scans of the Head and Neck Region
Brief Title: MRI-based Synthetic CT Images of the Head and Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: MRIguidance B.V. (Industry)
Responsible Party: Principal Investigator, Paul Merkus, Prof. Dr., Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022.0234; NL80426.029.22 (Registry Identifier: CCMO Register)
Record Dates: First submitted 2023-08-07; First posted 2023-08-29 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Imaging of Bony Structures of the Head (Various Conditions); Hearing Loss; Cholesteatoma; Sinusitis; Head and Neck Tumor
Keywords: MRI; Synthetic CT; Artificial Intelligence; Craniofacial
MeSH Terms: conditions — Hearing Loss; Cholesteatoma; Sinusitis; Head and Neck Neoplasms | interventions — Tomography, X-Ray Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: For all participants the same research activities will be performed (namely CT and MRI). The resulting paired MRI and CT scans will then be divided into a training set and a test set.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Other): Data from 25-35 participants will be used to train an algorithm to generate synthetic CT images from MRI scans.
  Interventions: Diagnostic Test: CT scan; Diagnostic Test: MRI scan
- Testing (Other): Data from remaining participants will be used to test the synthetic CT algorithm, by comparing true CT scans to synthetic CT scans made from MRI.
  Interventions: Diagnostic Test: CT scan; Diagnostic Test: MRI scan; Other: Synthetic CT scan

INTERVENTIONS:
Diagnostic Test: CT scan — Participants receive a CT scan of the head as part of their regular care. A larger part of the head will be scanned than for standard care.
Diagnostic Test: MRI scan — Participants receive an MRI scan, specifically for the purpose of the study.
Other: Synthetic CT scan — Synthetic CT scans will be generated from MRI scans, using the trained machine learning algorithm.
  Arms: Testing

SUMMARY:
In case of surgical procedures in the head and neck region, MRI in combination with CT of the bone is often the standard modality to visualise bony landmarks for planning, navigation and risk assessment. An important downside of a CT scan is the associated radiation exposure, especially in children. An additional downside is the sedation or general anaesthesia needed for both the MRI and CT scan session in very young children. These downsides could be removed if the CT scan can be substituted by an MRI sequence that can provide the same information as CT. This project aims to determine the feasibility of recreating CT like images of the craniofacial bones from MRI images using machine learning techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the outpatient ENT (Ear, Nose, Throat)-clinic.
* Aged 18 years or older.
* Referred for CT scan of the mastoid, sinonasal complex or face.

Exclusion Criteria:

* Pregnancy.
* Contra-indications for MRI or CT.
* Unwillingness to be informed about possibly clinically relevant, incidental findings from the MRI examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Geometrical accuracy. | Within one year after scans have been obtained.
  Geometrical accuracy of the bone morphology by determining the mean surface distance in mm between the cortical edges on synthetic CT and on true CT.
Radiodensity accuracy. | Within one year after scans have been obtained.
  Accuracy of the voxelwise radiodensity in Hounsfield Units and accuracy of the radiodensity contrast.
Visibility of landmarks. | Within one year after scans have been obtained.
  Accuracy of the visibility of clinically relevant anatomical landmarks on the synthetic CT images compared to the corresponding true CT images in the adult population, rated by experienced physicians on a 4-point Likert scale (1 = not visible, 4 = very well visible).

SECONDARY OUTCOMES:
Usefulness. | Within one year after scans have been obtained.
  Evaluation of potential usefulness of the synthetic CT images for surgical planning, surgical navigation and diagnostic purposes, as evaluated by experienced physicians and dichotomised into "useful" or "not useful".

CONTACTS AND LOCATIONS:
Overall Officials: Paul Merkus, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No